CLINICAL TRIAL: NCT05504174
Title: Detection of Circulating Tumor DNA Through Liquid Biopsies in Ovarian Cancer Patients and Evaluation of Prognostic and Predictive Values of Circulating Tumor DNA Assay.
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0698
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cell-free DNA extracted from frozen plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ovarian cancer group: Patients pathologically diagnosed with ovarian cancer
- Control group: Patients with benign or borderline adnexal mass

SUMMARY:
Ovarian cancer is the eighth most common cancer in women in Korea, with 2,600 cases occurring annually, and the number of cases is steadily increasing. There is no practical method for early detection of ovarian cancer, and 75 percent of patients are diagnosed with advanced stage. The treatment of ovarian cancer is based on surgical removal and platinum-based chemotherapy. The cell-free DNA (cfDNA) test has the advantage of being able to track and monitor mutations of tumor origin noninvasive.

The objective of this study was to assess the feasibility of circulating tumor DNA (ctDNA) as a biomarker for cancer recurrence in ovarian cancer after surgery. Diagnosis and prognosis evaluation using conventional methods such as CA-125, radiologic examination (CT), had limitations in diagnosing and prognostic observation of ovarian cancer. For precise diagnostic purposes, CA-125 had limitations because it was detected as positive value when the tumor size is enough large or states of metastasis, and CT-based diagnosis is practicable only when the size of tumor is detectable.

However, cell-free DNA can be detected even if the tumor size is small because it detects very small amount of mutation gene in the blood. In addition, the detection of tumor cell DNA from circulating blood can be a clinical decision making point whether to continue or stop chemotherapy.

In this study, the investigators collect whole blood from patients with ovarian cancer undergoing surgery. Control samples will be obtained from patients undergoing surgery for benign adnexal disease with CA125 >35U/ml. In ovarian cancer patients, blood samples will be collected prospectively every 3 months after surgery. Mutations found at the initial sample will be monitored during chemotherapy to investigate the ctDNA pattern. The primary outcome will be progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Female, over 19 years of age;
2. Patients with epithelial ovarian cancer
3. Patients with Serum CA-125 >35 U/mL

Exclusion Criteria:

1. Patients in pregnancy
2. Patients being treated for cancer of other organs, including gynecological cancer.
3. Patients who has difficulty reading and understanding Korean.
4. The tester's determination that the patient will not be able to comply with the clinical trial procedures.
5. Patients with severe infections or other serious medical problems that have resulted in impairment of the patient's function, making it difficult to the trial.

Ages: 19 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, with epithelial ovarian cancer and patients with benign adnexal disease with serum CA-125 >35 U/mL
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Determine Progression free survival (PFS) according to ctDNA pattern at time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Yun LEE, M.D., Principal Investigator — Department of Obstetrics and Gynecology, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No